CLINICAL TRIAL: NCT03179371
Title: Proteomic Analysis of Amniotic Fluid in the Case of Diaphragmatic Hernia: Search for Prognostic Expression Profiles
Brief Title: Proteomic Profiling for Congenital Diaphragmatic Hernia
Acronym: pro-CDH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: FEMTO-ST (Unknown)
Responsible Party: Sponsor
Other Study IDs: API/2016/78
Record Dates: First submitted 2017-05-16; First posted 2017-06-07 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Mothers whose fetus has CDH

SUMMARY:
Congenital diaphragmatic hernia (CDH) is a severe congenital malformation, related to a developmental defect of the diaphragm. The incidence of CDH is approximated at 1 in 3,000 live births. Although advances in surgery and neonatal intensive care have improved the prognosis, mortality remains high, around 30-50% related to severe lung hypoplasia and persistent pulmonary hypertension. Prenatal evaluation with observed/expected Lung over Head Ratio (o/e LHR), liver position and total lung volume measured by magnetic resonance, have been shown to correlate with neonatal mortality . However, the preponderant factor of persistent pulmonary hypertension remains difficult to predict prenatally. In patients with isolated diaphragmatic hernia (without associated malformations or karyotype abnormalities), prognosis is evaluated indirectly on pulmonary development from pulmonary volume measurements. Apart from the most caricatural cases with extremely good or very pejorative values, for a large proportion of fetuses with diaphragmatic dome hernia the prognosis remains uncertain.

The aim of the proposal is to investigate whether the analysis of the proteom of the amniotic fluid of the fetuses with CDH could give information of a prognostic character. The objective of the study is to identify, from the proteomic profile of the amniotic fluid of mothers whose fetus has CDH, prognostic markers candidates for death at 2 months of the infant. The first step is to carry out an exploratory and non-interventional study on a small sample (n = 10) of the target population. This is a preliminary step before considering, if the results are encouraging, a large-scale study from a biological collection to determine candidate proteins (new biomarkers) which relative expression levels could be used as surrogate marker of pulmonary hypoplasia.

DETAILED DESCRIPTION:
Pregnant patients for whom amniocentesis will be performed as part of the prenatal management of CDH confirmed by fetal ultrasound will be approached fot inclusion in the study. The indication of amniocentesis will be indicated according to the usual standards of care. Briefly, the study will not involve any additional invasive procedure. In our study, amniocentesis will be indicated during the conventional management of these patients. The needs of our research will not lead to additional amniocenteses, but simply an increase in the volume of amniotic fluid collected. An additional volume of 5 ml will be sampled for volumes usually taken from 20 to 30 ml. This volume of sampling will have a very limited impact on maternal and fetal well-being. An analysis of the proteom of the amniotic fluid of the patients will be carried out. The relative amounts of proteins and peptides contained in the amniotic fluid will be analyzed to explore variations in proteomic profile that may reflect different clinical gravity in terms of further evolution. The usual management of the patients and their children will not be modified by the procedures related to the research.

The first step will consist in carrying out a depletion of the major proteins, in particular albumin. A protein assay will be carried out from the same amount of protein for each sample (standardization). This depletion step will be followed by a migration step on a gel of 1D electrophoresis. Its purpose is both to eliminate all the contaminants that can hinder mass spectrometry analysis, to separate the proteins according to their molecular weight in order to simplify the protein mixture and to have a visual control of the heterogeneity of the sample. A differential visual analysis after staining will allow to define the highly variable zones between the groups of patients and within the same sample. We will select the zone of interest in identical manner for each sample and for the whole of the gel track. The use of commercial electrophoresis gels of the same batch and the parallel analysis of several samples of different groups and the use of quality controls ensure reproducibility. The proteins contained in these bands / gel zones are then digested according to a standardized protocol under controlled conditions. The simultaneous treatment of the different biological samples makes it possible to considerably reduce the impact of the variability of this step in the final differential statistical analysis. At the end of this step the proteins are analyzed by an LC-ESI MS / MS approach. This LC-ESI MS / MS approach consists of separating the peptides on a chromatographic separation column which is coupled directly to the ESI-MS / M mass spectrometer. This analytical approach can allow the identification of more than 1000 proteins and 5000 peptides. This analysis is repeated 3 times per sample so that analytical variability can be taken into account in differential statistical studies. At the end of this protocol the raw data of each zone are pooled by sample and the differential statistical study can be carried out.

ELIGIBILITY:
Inclusion Criteria:

Pregnant patients for whom amniocentesis will be performed as part of the prenatal diagnosis of a diaphragmatic hernia.

Exclusion Criteria:

* Refusal of patients,
* Refusal of spouse regarding data of the future child,
* Multiple malformations,
* Twin pregnancy,
* Prenatal diagnosis of an unconfirmed diaphragmatic hernia,
* Miscarriage after amniocentesis.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females
Study Population: Mothers whose fetus has CDH
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Neonatal death | 2 months of age

SECONDARY OUTCOMES:
Prenatal death of the fetus | 9 months
  Death during pregnancy
Neonatal death | 15 days
Apgar score | 5 min after birth
Age at surgery | 6 months of age
Need for a diaphragmatic prosthesis | 6 months of age
Duration of ventilation (in days) | 6 months of age
Duration of the oxygen dependency (in days) | 6 months of age
Need of supplemental oxygen therapy | 28 days of age
  Binary outcome (Yes/No)
Occurrence of pulmonary hypertension | 6 months of age
Duration of parenteral nutrition (in days) | 6 months of age
Age at the beginning of enteral nutrition | 6 months of age
Age at the beginning of oral nutrition | 6 months of age
Duration of hospital stay (in days) | 6 months of age

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - CHU de Dijon, Dijon

IPD SHARING:
Plan to Share IPD: No